CLINICAL TRIAL: NCT00285441
Title: Identification of Cytokine Profiles and T Cell Subsets Among Immunosuppressed Patients at Risk of Developing Active Tuberculosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Copenhagen Hospital Corporation (Other); The Danish Rheumatism Association (Other); Danish Lung Association (Other)
Other Study IDs: KF-01-278477
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2006-02-28 (Estimated); Status verified 2005-12

CONDITIONS: Tuberculosis; HIV Infections; Rheumatoid Arthritis
Keywords: HIV
MeSH Terms: conditions — Tuberculosis; HIV Infections; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to identify differences in TB specific immune responses among immunosuppressed patients latently infected with TB and patients with active TB.

DETAILED DESCRIPTION:
Immunosuppressed patients latently infected with TB are at higher risk of developing active TB than patients with normal immune functions. Especially two patient categories are at risk: HIV positives and patients receiving TNF-a blocking medication. Existing methods of diagnosis and surveillance of latent TB infection can not identify who will develop active TB and who can control the infection. There is a need for better understanding of TB specific immune functions,as we believe deficient TB specific immune reactions is a key in reactivation of latent TB infection.

In this study we follow groups of latent TB infected patients with either rheumatoid arthritis or HIV. We follow the patients during treatment with TNF-a blocking medication, HAART treatment or prophylactic TB medication. Results are correlated to patients with active TB, latent TB and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Latent TB infection + rheumatid arthritis
* Latent TB infection + HIV
* Active TB

Exclusion Criteria:

* Age < 18yrs
* Pregnancy
* Patients not able to understand the given information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-11; Study Completion 2008-09

CONTACTS AND LOCATIONS:
Overall Officials: Morten Ruhwald, MD, Principal Investigator — University Hospital Hvidovre
Locations (1):
- Infectious disease department University Hospital Hvidovre, Copenhagen, Denmark

REFERENCES:
- See also: Related Info — http://www.hvidovrehospital.dk